CLINICAL TRIAL: NCT06057753
Title: Personalized Video-based Education for Chronic Stroke Survivors: A Randomized Clinical Trial
Brief Title: MyStroke in Chronic Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Christopher Favilla, Assistant Professor of Neurology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 854145
Record Dates: First submitted 2023-08-22; First posted 2023-09-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Education (No Intervention): Standard stroke patient education as per the medical providers
- MyStroke (Experimental): Access to a personalized video-based stroke educational platform
  Interventions: Behavioral: MyStroke

INTERVENTIONS:
Behavioral: MyStroke — Personalized video-based stroke education platform
  Arms: MyStroke

SUMMARY:
This is a single-center randomized control trial assessing the impact of a personalized video-based educational platform on patients satisfaction and stroke knowledge in the context of chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. History of ischemic stroke between 1 and 10 years prior to enrollment
2. Receiving outpatient stroke care at the Hospital of the University of Pennsylvania
3. At least 18 years old
4. Access to a smart phone, tablet, or computer
5. Willingness to complete 2 follow-up surveys (7 days and 90 day post-enrollment)

Exclusion Criteria:

1. Unwilling or unable to access the customized app with a smartphone, tablet, or computer
2. Complete dependence on caregiver for all activities of daily living
3. Stroke occurred less than 1 year or greater than 10 years prior to screening/enrollment
4. Patient has severe aphasia (score of greater than or equal to 2 on National Institutes of Health Stroke Scale item 9)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with stroke education (90 days) | 90 days
  5-point Likert-scale (Q: I am satisfied with the quality of my stroke education; Answers range from strongly disagree to strongly agree)
Stroke etiology recognition (90 days) | 90 days
  The proportion of patients who correctly identify their stroke etiology
Stroke risk factor recognition (90 days) | 90 days
  The proportion of patients who correctly identify at least one of their vascular risk factors

SECONDARY OUTCOMES:
Stroke prevention medication recognition (7 days) | 7 days
  The proportion of patients who correctly identify their antithrombotic medications
Stroke prevention medication recognition (90 days) | 90 days
  The proportion of patients who correctly identify their antithrombotic medications
Patient satisfaction with stroke education (7 days) | 7 days
  5-point Likert-scale (Q: I am satisfied with the quality of my stroke education; Answers range from strongly disagree to strongly agree)
Stroke etiology recognition (7 days) | 7 days
  The proportion of patients who correctly identify their stroke etiology
Stroke risk factor recognition (7 days) | 7 days
  The proportion of patients who correctly identify at least one of their vascular risk factors
Stroke patient education retention (SPER) survey (7 days) | 7 days
  total score from the 5-question SPER (scale 0-10; higher score reflects better knowledge)
Stroke patient education retention (SPER) survey (90 days) | 90 days
  total score from the 5-question SPER (scale 0-10; higher score reflects better knowledge)
EuroQOL - visual analog scale (7 days) | 7 days
  patient-reported quality of life score (scale 0-100; higher score reflects better self-reported quality of life)
EuroQOL - visual analog scale (90 days) | 90 days
  patient-reported quality of life score (scale 0-100; higher score reflects better self-reported quality of life)
modified Rankin Scale | 90 days
  Ordinal functional disability scale (score 0 - 6)
Medication adherence (7 days) | 7 days
  total score of the Adherence Estimator (3 question survey; total score 0-36; higher score reflects higher risk of non-adherence)
Medication adherence (90 days) | 90 days
  total score of the Adherence Estimator (3 question survey; total score 0-36; higher score reflects higher risk of non-adherence)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States